CLINICAL TRIAL: NCT02031575
Title: Study on Mhealth and Reproductive Health in Teens
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: Weiss Family Program Fund for Research in Development Economics (Unknown); Harvard Lab for Economic Applications and Policy (Unknown)
Responsible Party: Principal Investigator, Slawa Rokicki, PhD Candidate, Harvard University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB13-1647
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Reproductive Health
Keywords: Reproductive Health; Contraception; Public Health; Sexual Health; Adolescents; Mobile Health

ARMS (3):
- Basic Treatment (Experimental): Sends messages to participants about reproductive health.
  Interventions: Behavioral: Basic Treatment
- Interactive Treatment (Experimental): Sends multiple choice questions and receives texts message responses from participants with incentive for responding correctly
  Interventions: Behavioral: Interactive Treatment
- Control (Placebo Comparator): Sends messages to students about malaria prevention and control.
  Interventions: Other: Control, comparator arm

INTERVENTIONS:
Behavioral: Interactive Treatment — Mobile phone text messaging service about reproductive health
  Arms: Interactive Treatment
Behavioral: Basic Treatment — Mobile phone text messaging service about reproductive health
  Arms: Basic Treatment
Other: Control, comparator arm
  Arms: Control

SUMMARY:
The purpose of the Study on Mhealth and Reproductive Health in Teens (SMART) is to evaluate the effectiveness of using text messages to improve the knowledge, communication, and attitudes about reproductive health among female adolescents in Greater Accra senior high schools. Previous research as well as qualitative work conducted by the Investigators shows that there are significant gaps in knowledge about reproductive health including on topics of pregnancy, sexually transmitted diseases, and contraception among secondary school students in Greater Accra. These gaps contribute to unwanted pregnancy and spread of sexually transmitted diseases. At the same time, phone ownership and use among young people has spread rapidly, especially in urban areas such as Accra. The Study on Mhealth and Reproductive Health (SMART) will seek to use mobile phone messages to increase awareness of these reproductive health issues among female adolescents in Accra. The objectives of SMART are to evaluate whether the messages can increase knowledge, increase communication, and improve attitudes towards reproductive health among adolescents in Greater Accra. By conducting a randomized controlled trial, we will be able to statistically evaluate if the messages have had any effect on improving outcomes for adolescents in the areas of knowledge, communication, and attitudes. This work can help guide future programs that can scale up this intervention and ultimately improve the health and wellbeing of adolescents across Ghana.

ELIGIBILITY:
Inclusion Criteria (for treated and control subjects):

* female
* aged 14-24
* secondary school student at day school

Exclusion Criteria (for treated and control subjects):

* male
* secondary school student at boarding school

Inclusion criteria (for spillover subjects):

* aged 14-24
* secondary school student at day school

Exclusion Criteria (for spillover subjects):

- secondary school student at boarding school

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1419 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Knowledge of Reproductive Health True/False Quiz of 20 questions | 5-6 months after baseline and then again 14-16 months after baseline
Sexual behavior | 14-16 months after baseline
  Assessed via a number of items: age at sexual debut, sex without a condom in the past year, pregnancy in the past year, ever had sex, use of condom at sexual debut, sex in the past year, used any contraception in the past year, used contraception at last sex, had an abortion

SECONDARY OUTCOMES:
Communication about reproductive health with family, friends, professional, and boyfriend | 3 months (asked 5-6 months after baseline and again 12-14 months after baseline)
  Communication is assessed via questionnaire items that ask the participant how often the participant has communicated with family, friends, professional, and boyfriend over the past 3 months.
Attitudes about reproductive health as measured by 5-point Likert type scale | 5-6 months after baseline and asked again 12-14 months after baseline
  Attitudes about reproductive health are measured via questionnaire items that ask participants about their attitudes about reproductive health. They respond via a 5-point Likert type scale.

OTHER OUTCOMES:
Spillover effect | 3-6 months
  Assess how much knowledge, communication, and attitudes spilled over to students in same school but not receiving any intervention
Process Measures | 3-6 months
  Assess whether students liked the intervention, whether they used it, and other questions designed to understand whether the mobile service was useful from students' perspectives
Heterogeneous effects | 3-6 months
  Assess whether treatment effects are heterogeneous along a number of dimensions: age (younger/older), category of school, and community connectedness.
Cost effectiveness | 3-6 months
  Assess whether the interactive treatment arm was cost effective compared to the basic treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Slawa Rokicki, MS, BS, Principal Investigator — Harvard University; Gunther Fink, PhD, Study Chair — Harvard School of Public Health (HSPH)
Locations (1):
- Innovations for Poverty Action, Accra, Greater Accra Region, Ghana

REFERENCES:
- [Derived] Rokicki S, Fink G. Assessing the reach and effectiveness of mHealth: evidence from a reproductive health program for adolescent girls in Ghana. BMC Public Health. 2017 Dec 20;17(1):969. doi: 10.1186/s12889-017-4939-7. PMID 29262823